CLINICAL TRIAL: NCT03903016
Title: A Randomized, Double-blind, Single-dose, 2-treatment, 2-period, 2-sequence Crossover Bioequivalence Study Comparing Two Different Strengths Formulations of Insulin Lispro Using the Euglycemic Clamp Technique, in Patients With Type 1 Diabetes Mellitus
Brief Title: A Bioequivalence Study Comparing Two Different Strengths Formulations of Insulin Lispro in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEQ15846; 2018-003131-30 (EudraCT Number); U1111-1207-8959 (Other: UTN)
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (T) (Experimental): Insulin Lispro (SAR342434), 200 Units/ml, single dose on day 1 of each period
  Interventions: Drug: Insulin Lispro SAR342434
- Reference (R) (Active Comparator): Insulin Lispro Sanofi® ,100 Units/ml, single dose on day 1 of each period
  Interventions: Drug: Insulin Lispro SAR342434

INTERVENTIONS:
Drug: Insulin Lispro SAR342434 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: Test (T)
Drug: Insulin Lispro SAR342434 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Other Names: Insulin lispro Sanofi®
  Arms: Reference (R)

SUMMARY:
Primary Objective:

To demonstrate bioequivalence between insulin lispro given as SAR342434, 200 Units/ml test formulation (T) and insulin lispro 100 Units/ml reference formulation (R) after a single subcutaneous (SC) dose

Secondary Objectives:

* To assess the pharmacodynamic profiles and further pharmacokinetic characteristics of the test formulation (T) in comparison to the reference formulation (R) after a single SC dose
* To assess the safety and tolerability of the test and the reference formulation of insulin lispro

DETAILED DESCRIPTION:
Study duration per participant is approximately 62 days including a screening period up to 28 days before first dose, 2 periods of 2 days, a wash out period of 5 to 18 days (preferred7 days) and an end of study visit 7 to 14 days after the last dose

ELIGIBILITY:
Inclusion criteria :

* Male or female patients, between 18 and 64 years of age, inclusive, with diabetes mellitus type 1 for more than one year
* Total insulin dose of <1.0 U/kg/day
* Fasting serum C-peptide <0.30 nmol/L at screening
* Glycohemoglobin (HbA1c) ≤75 mmol/mol (≤9%) at screening
* Stable insulin regimen for at least 2 months prior to study (day of insulin regimen switch, with respect to safety of the patient and scientific integrity of the study).
* Patients with anti-insulin antibody titer at screening ≤ 30.0 kU/L
* Body weight between 50.0 kg and 100.0 kg, inclusive, il male , and between 40.0 and 90.0 kg, inclusive, if female, Body Mass Index between 18 and 30.0 kg/m², inclusive

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness or any history or presence of HIT-type II (heparin induced thrombocytopenia Type II)
* More than 1 episode of severe hypoglycemia resulting in coma/seizures or requiring assistance of another person, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only, more than twice a month).
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* If female, pregnancy (defined as positive β-HCG blood test), breast-feeding

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetc (PK) parameter:INS-Cmax | 10 hours
  Maximum Insulin (INS) concentration
Assessment of PK parameter :INS-AUClast - | 10 hours
  Area under INS concentration time curve from 0 to last measurable concentration -

SECONDARY OUTCOMES:
Assessment of PK parameter:INS-AUC | 10 hours
  Area under INS concentration time curve from 0 to infinity
Assessment of PK parameter:INS-tmax | 10 hours
  Time to reach INS-Cmax
Assessment of PK parameter:INS-t1/2z | 10 hours
  INS terminal half life
Assessment of pharmacodynamic (PD) parameter:GIR-AUC0-8 | 8 hours
  Area under the Glucose Infusion Rate (GIR) time curve from 0 to 8 hours
Assessment of PD parameter:GIR-max | 8 hours
  Maximum smoothed GIR
Assessment of PD parameter:GIR-tmax | 8 hours
  Time to reach GIR-max
Duration of blood glucose control | 8 hours
  Duration of blood glucose control at or below 105 mg/dL
Adverse Events | Up to Day 62
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 2760001, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BEQ15846 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25219&tenant=MT_SNY_9011